CLINICAL TRIAL: NCT07035834
Title: SGLT-2 Inhibitors on Albuminuria in Chronic Kidney Disease Patients With Lupus Nephritis and ANCA- Associated Vasculitis: Study Design and Protocol
Brief Title: SGLT-2 Inhibitors on Albuminuria in Chronic Kidney Disease Patients With Lupus Nephritis and ANCA- Associated Vasculitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ivana Capuano, Researcher, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC001
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lupus Nephritis (LN); ANCA Associated Vasculitis (AAV)
Keywords: Lupus Nephritis; ANCA associated vasculitis; SGLT-2 inhibitors; nephroprotection
MeSH Terms: conditions — Lupus Nephritis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lupus nephritis and ANCA associated vasculitis patients treated with glifozines (Experimental)
  Interventions: Drug: Gliflozin

INTERVENTIONS:
Drug: Gliflozin — Our study will enroll non diabetic patients affected by chronic kidney disease secondary to lupus nephritis and ANCA associated vasculitis. Other studies have so far investigated only diabetic patients affected by the above mentioned diseases.

SUMMARY:
The goal of this clinical trial is to investigate the effect of the glifozines on albuminuria in chronic kidney disease patients affected by lupus nephritis and ANCA associated renal vasculitis. It will also learn about the safety of glifozines. The main questions it aims to answer are:

* Does glifozines lower the albuminuria of participants with chronic kidney disease secondary to lupus nephritis and ANCA associated renal vasculitis?
* What medical problems do participants have when taking glifozines?

Participants will:

* Take glifozines every day for 6 months.
* Baseline, 1 month and 6-month visits will be scheduled to collect demographic, clinical, biochemical, and urinary data.
* A psychosocial assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than18 years with chronic kidney disease from stage 1 to3, secondary to confirmed LN, without active LN, and AAV

Exclusion Criteria:

* 1) allergy or intolerance to SGLT2i exposure within 1month before screening; 2) recurrent urinary tract infections; 3) hepatic dysfunction (aspartate aminotransferase or alanine aminotransferase levels >2 times the upper normal limits); 4) an eGFR ˂30 ml/min/1.73 m2; 5) DM type I and II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The variation of albuminuria | From enrollment to the end of treatment at 6 months
The primary outcome is the variation of albuminuria after 6 months of treatment with SGLT-2i. | From enrollment to the end of treatment at 6 months

IPD SHARING:
Plan to Share IPD: No